CLINICAL TRIAL: NCT07285759
Title: Experimental Investigation of the Antibacterial Effect of Levobupivacaine on Staphylococcus Aureus in a Patient-Controlled Analgesia (PCA) Model
Brief Title: Investigation of Antibacterial Effect of Levobupivacaine on Staphylococcus Aureus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülay Akıncı, Dr. Gülay Akıncı, Department of Anesthesiology and Reanimation, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DEU-LEVOBUPI-2010; DEU-Anaesthesia-Study-2010 (Other: Dokuz Eylul University Faculty of Medicine)
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Staphylococcus Aureus Bacterial Contamination
Keywords: Levobupivacaine; Antibacterial effect; Patient Controlled Analgesia (PCA); Fentanyl; Scanning Electron Microscope (SEM); Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections | interventions — Levobupivacaine; Fentanyl; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Four independent groups were prepared using levobupivacaine and fentanyl at different concentrations and compared in parallel under in vitro laboratory conditions.
Masking Description: No masking was performed. The study was conducted as an open-label in vitro experimental model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - 0.125% Levobupivacaine + Fentanyl (Experimental): 0.125% levobupivacaine with 4 mL fentanyl (200 mcg) infused via PCA system for 24 hours.
  Interventions: Drug: Levobupivacaine; Drug: Fentanyl
- Group 2 - 0.0625% Levobupivacaine + Fentanyl (Experimental): 0.0625% levobupivacaine with 4 mL fentanyl (200 mcg) infused via PCA system for 24 hours.
  Interventions: Drug: Levobupivacaine; Drug: Fentanyl
- Group 3 - Fentanyl Only (Active Comparator): 4 mL fentanyl (200 mcg) infused via PCA system for 24 hours.
  Interventions: Drug: Fentanyl
- Group 4 - Saline (Control) (Placebo Comparator): 99 mL saline infused via PCA system for 24 hours.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Levobupivacaine — Levobupivacaine is a local anesthetic used at concentrations of 0.125% and 0.0625% to evaluate its antibacterial effect against Staphylococcus aureus in an in vitro PCA model.
  Arms: Group 1 - 0.125% Levobupivacaine + Fentanyl; Group 2 - 0.0625% Levobupivacaine + Fentanyl
Drug: Fentanyl — Fentanyl is an opioid analgesic used at a concentration of 200 mcg/4 mL, either alone or in combination with levobupivacaine, to assess potential contribution to antibacterial activity.
  Arms: Group 1 - 0.125% Levobupivacaine + Fentanyl; Group 2 - 0.0625% Levobupivacaine + Fentanyl; Group 3 - Fentanyl Only
Other: Saline — Sterile saline solution (99 mL) used as the control group to compare antibacterial activity in the PCA infusion model.
  Arms: Group 4 - Saline (Control)

SUMMARY:
This experimental in vitro study aimed to investigate the antibacterial effect of levobupivacaine on Staphylococcus aureus in a patient-controlled analgesia (PCA) model at concentrations commonly used for postoperative pain treatment (0.125%) and painless labour (0.0625%). The antibacterial activity was evaluated using colony count reduction and supported by Scanning Electron Microscope (SEM) imaging.

DETAILED DESCRIPTION:
Study solutions were prepared as 100 mL each. Four groups were designed:

* Group 1: 0.125% levobupivacaine + 4 mL fentanyl (200 mcg)
* Group 2: 0.0625% levobupivacaine + 4 mL fentanyl (200 mcg)
* Group 3: 4 mL fentanyl (200 mcg)
* Group 4: 99 mL saline (control)

Each group received 1 mL of Staphylococcus aureus 0.5 McF (1.5×10⁸ cfu/mL). All samples were infused through a Portex bacterial filter at 4 mL/h for 24 hours using PCA devices. Samples collected from bottles, filter inlets, and outlets were cultivated on Blood Agar. Colony counts were compared statistically using the Kruskal-Wallis and Mann-Whitney U tests (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Laboratory study using Staphylococcus aureus bacterial cultures.
* Samples exposed to different concentrations of levobupivacaine and fentanyl solutions.
* Controlled laboratory environment (Dokuz Eylül University, Microbiology Laboratory).

Exclusion Criteria:

* No human participants included.
* No animal models used.
* Studies outside the defined experimental conditions were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Reduction in Staphylococcus aureus Colony Count | 24 hours
  Quantitative measurement of the antibacterial effect of levobupivacaine and fentanyl by counting Staphylococcus aureus colonies grown on Blood Agar after 24-hour PCA infusion at different concentrations.

SECONDARY OUTCOMES:
Morphological Changes of Staphylococcus aureus under SEM | 48
  Evaluation of ultrastructural changes in Staphylococcus aureus cells after exposure to levobupivacaine and fentanyl using Scanning Electron Microscope (SEM) imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Akıncı, Principal Investigator — Dokuz Eylul University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study was completed in 2011 and data sharing was not included in the original ethics approval.

REFERENCES:
- See also: Related Info — https://debis.deu.edu.tr/